CLINICAL TRIAL: NCT07114614
Title: Fatty Acid Binding Proteins and Markers of Cellular Senescence in Cancer Survivors
Status: Not yet recruiting | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: CASE5Z25
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Marker; Structural
Keywords: Fatty Acid Binding Proteins; Cancer Survivors; FABP4 and FABP5

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer participants
  Interventions: Other: Specimen #1; Other: Specimen #2
- Control Group
  Interventions: Other: Specimen #1; Other: Specimen #2

INTERVENTIONS:
Other: Specimen #1 — Specimen 1 will be collected in a 10 ml SST (serum separator tube).
Other: Specimen #2 — Specimen #2 will be collected in a 10 ml SST (serum separator tube)

SUMMARY:
The purpose of this research study is to investigate whether cancer survivors have higher levels of proteins called Fatty Acid Binding Proteins as well as 12 different markers of cellular senescence than people who have never had cancer. Investigators believe that these levels may be elevated in cancer survivors as a result of their cancer and the treatments they received and may put them at higher risk for chronic conditions such as high cholesterol, diabetes, high blood pressure, and obesity. This study will also compare the levels of these proteins and inflammatory markers in the blood with different aspects of cancer treatment the survivors received. Investigators are investigating if there is a correlation between levels of these proteins and markers, the type of treatment cancer survivors received, and development of metabolic conditions.

DETAILED DESCRIPTION:
Recent advances in cancer-directed therapies for pediatric patients has led to increasing numbers of survivors of childhood and young adult cancers who face unique long term health risks as a result of their cancer and the exposure to tissue damaging agents, including chemotherapy, radiation therapy and immune modulating agents. Risks associated are often dependent on the type of cancer, age at diagnosis, and treatment received with many agent-specific potential late effects . However, previous studies of childhood and young adult cancer survivors have shown that they are at significantly increased risk for metabolic late effects including obesity, hypertension, dyslipidemia, diabetes and insulin resistance, and cardiovascular disease. These risks have been shown to be even higher for survivors treated with specific therapies such as abdominal or total body irradiation and for those treated at a younger age . Proposed mechanisms of increased risk of metabolic late effects include alterations to the hypothalamic-pituitary-adrenal axis, pancreatic insufficiency, changes in leptin and adiponectin signaling, disturbances in signaling due to sarcopenic obesity, poor dietary and exercise habits, and treatment-induced changes to the gut microbiome . Population-based studies have shown that survivors of childhood cancers are at significantly higher risks than their siblings for cardiovascular events, insulin resistance, hypertension, and obesity and this risk is increased for survivors who were obese at diagnosis and who had significant increase in body mass index (BMI) compared to prior to diagnosis. However, a mechanism that explains why survivors of childhood and young adult cancers are at significantly increased risk of chronic metabolic disease compared to their siblings has not yet been elucidated. Though studies examining the effect of diet and exercise programs for childhood cancer survivors at risk for chronic metabolic disease have shown significant risk reduction, survivors remain at significant risk for early morbidity and mortality from metabolic late effects.

Fatty Acid Binding Proteins (FABPs) are a group of intracellular lipid chaperones that bind hydrophobic molecules and traffic them to different organelles, supporting cellular functions such as oxidation for energy, cell membrane synthesis, and transcription regulation. Though FABPs are found in many different organs throughout the body and serve organ-specific functions, FABP4 and FABP5 have been found to have specific roles in obesity and metabolic disease. FABP4 is found in highest concentrations in adipose tissue, though is also found in macrophages, and is thought to play a role in obesity-associated chronic inflammation. FABP5 is found in highest concentrations in macrophages and has been demonstrated to play a significant role in development of cardiovascular disease. In addition to their role in chronic metabolic diseases, FABPs have been shown to play a role in cancer metastasis, resistance to treatment, and tumor recurrence. A recent study in Poland examined levels of FABP4 and FABP5 in association with metabolic syndrome in survivors of childhood Acute Lymphoblastic Leukemia (ALL), finding that levels of FABP4 were significantly elevated in survivors of childhood ALL compared to controls, but to investigator's knowledge no other studies have examined the association of FABPs and metabolic late effects in survivors of childhood and young adult cancers.

In addition to being at increased risk for metabolic diseases, survivors of childhood and young adult cancers have been described as having an accelerated aging phenotype associated with early onset of osteopenia and osteoporosis as well as frailty. One hypothesis for the underlying mechanism for this accelerated aging phenotype is induction of cellular senescence by cancer-directed therapies. The number of senescent cells increases with age and has been associated with many different age-related diseases, thought to be due to a combination of DNA damage, protein misfolding, and peroxidation on the cellular level leading to growth arrest and eventual cell death. The Senescence Associated Secretory Phenotype (SASP) has been described and attempts have been made to identify reliable biomarkers to predict who is at risk for senescence-associated diseases as well as targets for senolytic therapies to reduce risk. While chemotherapeutic agents and radiation use distinct mechanisms to interrupt cancer cell replication and viability, they concomitantly impact the health of normal cells repeatedly exposed to these agents in the process of cancer therapy. This has been demonstrated in mouse models when circulating SASP biomarkers were found to be elevated after mice were exposed to chemotherapeutic agents; levels of these markers correlated in women undergoing breast cancer treatment with more severe chemotherapy side effects such as neuropathy, nausea, and low blood counts. Some SASP markers have been demonstrated to be predictive of post-surgical outcomes, but have not been examined in survivors of childhood and young adult cancers .

Though population-based studies have shown significant increased risk for early development of metabolic diseases such as dyslipidemia, hypertension, insulin resistance, cardiovascular disease, and obesity in survivors of childhood and young adult cancers, the underlying cellular mechanisms remain incompletely described. Additionally, reliable biomarkers predicting risk of adverse outcomes in survivor populations have not been established. This study aims to determine whether circulating FABPs 4/5 and SASP biomarkers are elevated in survivors of childhood and young adult cancers compared to healthy controls, potentially providing information to help determine who is most at risk for chronic metabolic effects of cancer therapy and eventually serving as therapeutic targets to combat metabolic late effects of cancer and cancer-directed therapies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of at least one malignancy for which chemotherapy, radiation, and/or stem cell transplantation was utilized as part of treatment
* Completed all therapeutic interventions for their malignancy and are at least 2 years off therapy
* At least 1-year post-stem cell transplant for malignant condition

Exclusion Criteria:

1. Pregnancy at the time of the study
2. Any autoimmune condition including but not limited to lupus, rheumatoid arthritis, Crohn's disease, ulcerative colitis, type 1 diabetes, EXCEPT well-controlled autoimmune hypothyroidism for at least 6 months
3. Presence of active graft versus host disease
4. Malignancy treated using surgery only
5. Acute relapsed disease or second malignancy
6. Transplant for non-malignant conditions (e.g. cell disease, Hurler syndrome)
7. Currently taking systemic steroids and/or immunosuppressant medications
8. Acute illness necessitating hospitalization in the 30 days prior to blood draw
9. Presence of a chronic inflammatory disease EXCEPT obesity
10. Fever, active infection or inflammation, or taking antibiotics at the time of blood draw
11. A diagnosis of Type 2 diabetes or Hypertension treated with medication
12. Currently lipid lowering medications
13. Growth hormone deficiency or hypothalamic dysfunction

Ages: 5 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: For pediatric control participants, labs will be drawn with IV placement prior to procedure or sedation. Measurements will be taken during the same visit. If desired by patient and parent, a separate research visit can be arranged for participants to have labs drawn at their convenience.
  For adult control participants, a research visit will be arranged at the participants' convenience for measurements to be obtained and study labs to be drawn.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Correlation between FABP levels and the development of risk factors for metabolic syndrome and inflammation | Baseline
To determine the correlation with types of cancer-directed therapy received. | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Case Comprehensive Cancer Center, UH Rainbow Babies & Children's Hospital, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No